CLINICAL TRIAL: NCT05623423
Title: Evaluation of Clinical Performance of Class IV Restoration Using Organically Modified Ceramic (OMNOCER) in Comparison to a Methacrylate Based Composite Resin a Randomized Clinical Trial
Brief Title: Evaluation of Clinical Performance of Class IV Restoration Using Organically Modified Ceramic (OMNOCER) in Comparison to a Methacrylate Based Composite Resin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lilly Assem Mousa Ahmed, Investigator, data entry & corresponding author B.D.S. October University for Modern Sciences and Arts (2017). Teaching Assistant at MSA University, 6th Of October, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: class IV restoration
Record Dates: First submitted 2022-11-06; First posted 2022-11-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2022-12

CONDITIONS: Shade Match
Keywords: class IV restoration; ORMOCER; methacrylate based composite resin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organically Modified Ceramic (ORMOCER) Resin Composite. (Experimental): (Admira Fusion, Voco GmbH, Germany)
  Interventions: Other: (Admira Fusion, Voco GmbH, Germany)
- Methacrylate Based Composite (Active Comparator): (Ceram.X Spectra ST, Dentsply Sirona, UK)
  Interventions: Other: Methacrylate Based Composite

INTERVENTIONS:
Other: (Admira Fusion, Voco GmbH, Germany) — cavity margins will be extended to the proximal area, incisal edge, facial and lingual surfaces All enamel margins will be beveled at a 45° angle to the external cavosurface.(approximately 0.5-2.0 mm) An impression for the upper anterior teeth will be taken to produce a silicon palatal index The proximal margins of the restorations will be achieved using the Unica anterior matrix teeth will be etched using 37% phosphoric acid gel for 30 s then rinsed with air water for 20 s A single coat of universal bond cured using and LED light curing unit for 10 s Using the chosen enamel shade of the ORMOCER Resin Composite a thin layer (0.5-1 mm) Unica matrix will used to produce the proximal margins of the restorations Contouring, finishing and polishing of the restoration will be done Dental floss and finishing strips will be used Rubber dam will then be removed and occlusion will be checked using an articulating paper
  Arms: Organically Modified Ceramic (ORMOCER) Resin Composite.
Other: Methacrylate Based Composite — The exact same steps as in the intervention will be done but using the chosen shades of Methacrylate Based Composite Resin. (Ceram.X Spectra ST, Dentsply Sirona, UK)
  Arms: Methacrylate Based Composite

SUMMARY:
Evaluation of clinical performance of class IV restoration using organically modified ceramic (ORMOCER) in comparison to a Methacrylate Based Composite Resin: A randomized clinical trial

DETAILED DESCRIPTION:
Statement of the problem:

Resin composites have been the most popular material in esthetic dentistry since 1960's. Esthetic restorative material should resemble the natural tooth; in both color match and stability, and should have adequate strength, wear and sealing characteristics

. Longevity of anterior restorations varied in earlier studies depending on the restorative material and cavity class. Involvement of the incisal angle in anterior teeth resulted in accompanied reduction in average survival time. In contrast to class I, II, III and V cavity configurations, class IV restorations are stressed at the incisal angle, posing a challenge to the tooth restoration interface. Because the majority of class IV restorations lack mechanical retention; the tooth-bonded interface faces additional obstacles. In addition, color is one of the most important factors of esthetic restorations, since color change may be due to intrinsic factors as; changes in the filler, matrix and silane coating as well as extrinsic staining; as absorption of stains, chemical reactivity, diet and oral hygiene. But the recent advances in the resin composite restoration in their monomer chemistry, filler type and structure have been continuously developed to improve their mechanical and physical properties.

Rationale:

In order to optimize the properties of the material and facilitate deeper light transmission, manufacturers incorporated an advanced composite filler technology and resin matrix modifications by introducing Organically Modified Ceramics with pure silicate technology showing superior material properties, which was claimed to be better than Methacrylate Based Composite Resin. Moreover, polymerization shrinkage stresses depend on many factors, like composition of resin matrix, quantity of filler and degree of conversion. Ormocer induces polymerization as a result of a matrix of long inorganic silica chains with organic lateral chains. This type of Ormocer enhances aesthetics, color stability, abrasion resistance, and reduces polymerization shrinkage and surface roughness due to the presence of ceramic polysiloxane, which has low degree of polymerization shrinkage (1.25%)

ELIGIBILITY:
Inclusion Criteria:

participant:

1. Age of patient (18-40) years old.
2. Good oral hygiene.

Teeth:

1. Having no active pulpal or periodontal conditions.
2. Normal Occlusion.
3. Able to return for follow-up assessments as illustrated by the examiners. -

Exclusion Criteria:

participant:

1. Patients with Edge-to-Edge occlusion.
2. Patients with high caries index.
3. Patients with uncontrolled para-functional habits (e.g. bruxism or clenching).
4. Patients with inadequate oral hygiene.
5. Patients with periodontal or gingival conditions.
6. Patients with orthodontic appliances.
7. Patients with spontaneous pain or sensitivity to percussion
8. Pregnant Patients -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Shade match | T1: 1 week (baseline)
  measured by Modified USPHS
Shade match | T2: 3 months
  measured by Modified USPHS
Shade match | T3: 1 year.
  measured by Modified USPHS

SECONDARY OUTCOMES:
a) Retention rate | T1: 1 week (baseline)
  Modified united states public health service
a) Retention rate | T2: 3 months
  Modified united states public health service
a) Retention rate | T3: 1 year
  Modified united states public health service

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Abdulhameed, Professor, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Barcellos DC, Batista GR, Silva MA, Pleffken PR, Rangel PM, Fernandes VV Jr, Di Nicolo R, Torres CR. Two-year clinical performance of self-etching adhesive systems in composite restorations of anterior teeth. Oper Dent. 2013 May-Jun;38(3):258-66. doi: 10.2341/11-397-C. Epub 2012 Oct 30. PMID 23110580
- [Background] Blum SL, Horn M, Olms C. A comparison of intraoral spectrophotometers-Are there user-specific differences? J Esthet Restor Dent. 2018 Sep;30(5):442-448. doi: 10.1111/jerd.12407. Epub 2018 Aug 25. PMID 30144376
- [Background] Cetin AR, Unlu N, Cobanoglu N. A five-year clinical evaluation of direct nanofilled and indirect composite resin restorations in posterior teeth. Oper Dent. 2013 Mar-Apr;38(2):E1-11. doi: 10.2341/12-160-C. Epub 2012 Dec 5. PMID 23215545
- [Background] Demirci M, Tuncer S, Sancakli HS, Tekce N, Baydemir C. Five-year Clinical Evaluation of a Nanofilled and a Nanohybrid Composite in Class IV Cavities. Oper Dent. 2018 May/Jun;43(3):261-271. doi: 10.2341/16-358-C. Epub 2018 Mar 13. PMID 29533716
- [Background] Frese C, Wohlrab T, Soliman S, Hahn B, Busch C, Babai A, Krastl G, Wolff D. A Multicenter Trial on the Long-term Performance of Direct Composite Buildups in the Anterior Dentition - Survival and Quality Outcome. J Adhes Dent. 2020;22(6):573-580. doi: 10.3290/j.jad.a45514. PMID 33491402
- [Background] Gresnigt MM, Kalk W, Ozcan M. Randomized controlled split-mouth clinical trial of direct laminate veneers with two micro-hybrid resin composites. J Dent. 2012 Sep;40(9):766-75. doi: 10.1016/j.jdent.2012.05.010. Epub 2012 Jun 2. PMID 22664565
- [Background] Karaman E, Yazici AR, Ozgunaltay G, Ustunkol I, Berber A. Clinical Evaluation of a Silorane- and a Methacrylate-Based Resin Composite in Class II Restorations: 24-Month Results. Oper Dent. 2017 Jul/Aug;42(4):E102-E110. doi: 10.2341/15-286-C. PMID 28682704
- [Background] Llena C, Fernandez S, Forner L. Color stability of nanohybrid resin-based composites, ormocers and compomers. Clin Oral Investig. 2017 May;21(4):1071-1077. doi: 10.1007/s00784-016-1850-z. Epub 2016 May 16. PMID 27183827
- [Background] Rajeev V, Arunachalam R, Nayar S, Arunima PR, Ganapathy S, Vedam V. "Ormocer an innovative technology": A replacement for conventional cements and veneer? A comparative in vitro analysis. Eur J Dent. 2017 Jan-Mar;11(1):58-63. doi: 10.4103/ejd.ejd_113_16. PMID 28435367
- [Background] Ribeiro JS, Peralta SL, Salgado VE, Lund RG. In situ evaluation of color stability and hardness' decrease of resin-based composites. J Esthet Restor Dent. 2017 Sep;29(5):356-361. doi: 10.1111/jerd.12319. Epub 2017 Jul 24. PMID 28737281
- [Background] Romero MF, Haddock FJ, Freites AG, Brackett WW, Brackett MG. Restorative Technique Selection in Class IV Direct Composite Restorations: A Simplified Method. Oper Dent. 2016 May-Jun;41(3):243-8. doi: 10.2341/15-158-T. Epub 2016 Feb 26. PMID 26919082
- [Background] Ruschel VC, Martins MV, Bernardon JK, Maia HP. Color Match Between Composite Resin and Tooth Remnant in Class IV Restorations: A Case Series. Oper Dent. 2018 Sep/Oct;43(5):460-466. doi: 10.2341/17-132-S. Epub 2018 Mar 16. PMID 29547347
- [Background] Sebold M, Lins RBE, Sahadi BO, Santi MR, Martins LRM, Giannini M. Microtensile Bond Strength, Bonding Interface Morphology, Adhesive Resin Infiltration, and Marginal Adaptation of Bulk-fill Composites Placed Using Different Adhesives. J Adhes Dent. 2021 Oct 1;23(5):409-420. doi: 10.3290/j.jad.b2000221. PMID 34549924
- [Background] Torres C, Augusto MG, Mathias-Santamaria IF, Di Nicolo R, Borges AB. Pure Ormocer vs Methacrylate Composites on Posterior Teeth: A Double-blinded Randomized Clinical Trial. Oper Dent. 2020 Jul 1;45(4):359-367. doi: 10.2341/19-079-C. PMID 32053457
- [Background] van Dijken JW, Pallesen U. Fracture frequency and longevity of fractured resin composite, polyacid-modified resin composite, and resin-modified glass ionomer cement class IV restorations: an up to 14 years of follow-up. Clin Oral Investig. 2010 Apr;14(2):217-22. doi: 10.1007/s00784-009-0287-z. Epub 2009 Jun 6. PMID 19504133